CLINICAL TRIAL: NCT01871272
Title: Knee Arthroscopy Cohort Southern Denmark (KACS)
Acronym: KACS
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Lillebaelt Hospital, Kolding and Vejle, Denmark (Unknown)
Responsible Party: Principal Investigator, Jonas Bloch Thorlund, Associate Professor, University of Southern Denmark
Other Study IDs: 2012-41-1411; #12-125457 (Other Grant/Funding Number: The Danish Council for Independent Research | Medical Sciences); #12/6334 (Other Grant/Funding Number: Region of Southern Denmark)
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Meniscus Injury; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Meniscus Injury Patients: Patients having surgery for a meniscal tear.
  Interventions: Procedure: Arthroscopic Meniscus Surgery

INTERVENTIONS:
Procedure: Arthroscopic Meniscus Surgery — Surgery to the meniscus - resection or repair.

SUMMARY:
PURPOSE: To investigate the natural time course of patient-reported outcomes after meniscus surgery and identify factors associated with good and bad outcome after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Assigned for arthroscopy on suspicion of a medial and/or lateral meniscus tear.
* Age >18 years at time of recruitment
* Having an email address
* Able to read and understand Danish

Exclusion Criteria:

* Patients who will or have previously undergone surgical reconstruction of the anterior or posterior cruciate ligament (ACL or PCL) in either knee
* Fracture to the lower extremities (i.e. hip, leg or foot) in either leg within the last 6 months prior to recruitment
* Not mentally able to reply to the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assigned for arthroscopy on suspicion of a meniscus tear in the period from February 1st 2013 to January 31st 2014 will be consecutively recruited to the KACS cohort from 4 different hospitals (Lillebaelt Hospital - Kolding and Vejle and Odense University Hospital - Odense and Svendborg) in the Region of Southern Denmark.
Sampling Method: Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | PRE surgery (assessed 1-14 days prior to surgery) and at 12 weeks and 52 weeks follow-up
  Knee specific questionnaire. All domains on the KOOS. Primary end point is change from PRE surgery (assessed 1-14 days prior to surgery) to 52 weeks follow-up.

SECONDARY OUTCOMES:
Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) | PRE surgery (assessed 1-14 days prior to surgery) and at 12 weeks and 52 weeks follow-up.
  Generic health survey questionnaire.
Patient Acceptable Symptom State (PASS) | At 12 weeks and 52 weeks follow-up.
  Dichotomous outcome (y/n) to the question: "Considering your knee function, do you feel that your current state is satisfactory? With knee function you should take into account all activities you have during your daily life, sport and recreational activities, your level of pain and other symptoms, and also your knee related quality of life".
Treatment failure (TF) | At 12 weeks and 52 weeks follow-up.
  Patients replying "no" to the PASS question will also be asked to answer (y/n) the following question: "Would you consider your current state as being so unsatisfactory that you think the treatment has failed?". Patients replying, "yes" to the second question will be defined as experiencing "treatment failure" (TF).

OTHER OUTCOMES:
Global perceived effect (GPE) | At 12 weeks and 52 weeks follow-up.
  Questions regarding global perceived effect (GPE) to explore minimal clinical important change in patient-reported outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas B Thorlund, PhD, Principal Investigator — Department of Sports Science and Clinical Biomechanics, University of Southern Denmark
Locations (4):
- Denmark (4):
  - Department of Orthopedics, Lillebaelt Hospital, Kolding, Southern Denmark
  - Department of Orthopedics and Traumatology, Odense University Hospital, Odense, Southern Denmark
  - Department of Orthopedics and Traumatology, Odense University Hospital, Svendborg, Southern Denmark
  - Department of Orthopedics, Lillebaelt Hospital, Vejle, Southern Denmark

REFERENCES:
- [Background] Thorlund JB, Christensen R, Nissen N, Jorgensen U, Schjerning J, Porneki JC, Englund M, Lohmander LS. Knee Arthroscopy Cohort Southern Denmark (KACS): protocol for a prospective cohort study. BMJ Open. 2013 Oct 14;3(10):e003399. doi: 10.1136/bmjopen-2013-003399. PMID 24127057
- [Derived] Giladi JO, Holsgaard-Larsen A, Varnum C, Thorlund JB. Sports Participation and Performance 5 Years After Arthroscopic Partial Meniscectomy: A Retrospective Cohort Study of 288 Patients. J Orthop Sports Phys Ther. 2022 Apr;52(4):224-232. doi: 10.2519/jospt.2022.10785. PMID 35442751
- [Derived] Pihl K, Ensor J, Peat G, Englund M, Lohmander S, Jorgensen U, Nissen N, Fristed JV, Thorlund JB. Wild goose chase - no predictable patient subgroups benefit from meniscal surgery: patient-reported outcomes of 641 patients 1 year after surgery. Br J Sports Med. 2020 Jan;54(1):13-22. doi: 10.1136/bjsports-2018-100321. Epub 2019 Jun 11. PMID 31186258
- [Derived] Thorlund JB, Pihl K, Nissen N, Jorgensen U, Fristed JV, Lohmander LS, Englund M. Conundrum of mechanical knee symptoms: signifying feature of a meniscal tear? Br J Sports Med. 2019 Mar;53(5):299-303. doi: 10.1136/bjsports-2018-099431. Epub 2018 Aug 31. PMID 30170997
- [Derived] Thorlund JB, Englund M, Christensen R, Nissen N, Pihl K, Jorgensen U, Schjerning J, Lohmander LS. Patient reported outcomes in patients undergoing arthroscopic partial meniscectomy for traumatic or degenerative meniscal tears: comparative prospective cohort study. BMJ. 2017 Feb 2;356:j356. doi: 10.1136/bmj.j356. PMID 28153861